CLINICAL TRIAL: NCT01981369
Title: Effect of Intravenous Dexmedetomidine on the Analgesic Duration of Infraclavicular Block With Ropivacaine for Upper Limb Surgery: a Prospective, Randomized, Double Blind Study
Brief Title: Effect of Intravenous Dexmedetomidine on Analgesic Duration of Infraclavicular Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Shalini Dhir, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 104572
Record Dates: First submitted 2013-11-05; First posted 2013-11-11 (Estimated); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Postoperative Pain
Keywords: Dexmedetomidine sedation; Regional Anesthesia; Infraclavicular block
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propofol sedation. (Active Comparator): This group will have infraclavicular block and sedation during surgery with intravenous Propofol. Patients will receive intravenous Propofol sedation 50-100 mcg/kg/min infusion. The infusion will be stopped 15 minutes before the end of surgery.
  Interventions: Drug: Propofol; Procedure: Infraclavicular block
- Dexmedetomidine sedation. (Experimental): This group will have infraclavicular block and sedation with intravenous Dexmedetomidine. Patients will receive intravenous Dexmedetomidine sedation bolus 0.5mcg/kg in 10 minutes and then 0.2-0.5 mg/kg/hr infusion. The infusion will be stopped 15 minutes before the end of surgery.
  Interventions: Drug: Dexmedetomidine; Procedure: Infraclavicular block

INTERVENTIONS:
Drug: Dexmedetomidine — Intravenous sedation with dexmedetomidine
  Other Names: Precedex
  Arms: Dexmedetomidine sedation.
Drug: Propofol — Intravenous sedation with propofol
  Arms: Propofol sedation.
Procedure: Infraclavicular block — All patients will receive ultrasound guided infraclavicular block with the standard protocol of the Block Room in St. Joseph Hospital.

SUMMARY:
The study will evaluate the effect of Dexmedetomidine sedation on the duration of infraclavicular block in patients scheduled for surgery of elbow, forearm and/or hand. All patients will receive infraclavicular block before the surgery and then they will be randomized to receive either Dexmedetomidine or Propofol sedation. Duration of the sensory block will be evaluated in recovery room, 24 and 48 hours after the surgery.

Hypothesis:

Primary: Dexmedetomidine sedation increases the duration of sensory infraclavicular block in patients scheduled for upper limb surgery.

Secondary: Dexmedetomidine sedation

* Gives an adequate level of sedation during the surgical procedure
* Reduces the requirements of postoperative opioids
* Improves the quality of sleep on the night of the surgery
* Increases patients satisfaction regarding the anesthesia technique
* Dexmedetomidine sedation is safe and easy to use
* Dexmedetomidine sedation provides less respiratory depression during the procedure.

DETAILED DESCRIPTION:
Methodology:

Study design A randomized, prospective, double blind study.

Patient groups Group 1 (control group) This group will have infraclavicular block and sedation during surgery with intravenous Propofol.

Group 2 (intervention group) This group will have infraclavicular block and sedation with intravenous Dexmedetomidine.

Recruitment and Informed consent: Recruitment will take place in the preoperative clinic or surgical day care unit.

Duration of study: We estimate that 3 patients per week will be eligible and agree to participate. One year should therefore provide adequate time for study completion.

Data analysis:

Descriptive statistics will be used to present baseline characteristics for the two groups.

T-test or Mann-Whitney U- test will be used to compare these baseline values between the two groups. Quantitative data like pain scores and narcotic consumption will be compared using repeated measures ANOVA within the groups and two tailed unpaired t-test between groups (or Mann- Whitney-U test if skewed distribution). The nonparametric data will be analyzed using Chi squared test. P less than 0.05 will be considered statistically significant. Continuous variables will be assessed for normality and will be presented as mean (SD) or median with interquartile range (IQR) as appropriate. Categorical variables will be assessed using frequency tables and Fisher's exact test. The interval between the onset of the sensory block and first analgesic request will be analyzed by Kaplan-Meier survival analysis.

Protocol: The study will be performed on patients undergoing ambulatory hand, forearm or elbow surgery. After informed consent, the patients will be randomized to a study group using a computer generated random number table and sealed envelope technique. Following this the patients will be taken to the block room for performing the infraclavicular block, using standard monitors that will include non-invasive blood pressure, electrocardiogram and pulse oximetry.

All patients will receive ultrasound guided infraclavicular block with the standard protocol of the Block Room in St. Joseph Hospital. After the block, the patient will be moved to the operating room for the surgery where sedation with Dexmedetomidine or Propofol will be started as per the randomization. In order to blind the patient, the syringe and tubing will be covered with towels. The patients will be allocated to one of the two groups:

Group 1: Patients will receive intravenous Dexmedetomidine sedation bolus 0.5mcg/kg in 10 minutes and then 0.2-0.5 mg/kg/hr infusion. The infusion will be stopped 15 minutes before the end of surgery.

Group 2: Patients will receive intravenous Propofol sedation 50-100 mcg/kg/min infusion. The infusion will be stopped 15 minutes before the end of surgery.

Sedation score and hemodynamic profile during the surgery will be recorded every 15 minutes. Oxygen will be provided through facial mask. Total dose of narcotic used will be recorded.

After the surgical procedure, patients will be moved to the Post Anesthetic Care Unit (PACU), where an independent blinded observer not involved in the performance of the block or intraoperative care of the patient, will follow up the patients in the postoperative period.

The patients will be assessed for the site and severity of pain at rest at the arrival in the PACU. Pain score will be the Numerical Rating Score (NRS) on a scale of 0 to 10 where 0 is no pain and 10 the worst pain ever experienced. Data regarding duration of surgery and the duration of stay in PACU will also be collected from the nursing records. Opioids requirement in PACU will also be collected from these records. Complications, if any will be noted.

The patients will be assessed for pain at the surgical site at the time of discharge from PACU. They will also be given a diary to take home. Patient will be educated regarding the NRS and asked to record in the diary after discharge from the PACU until 20:00 hours. They will also be asked to record when they require first analgesic dose, the time of return of sensation in dorsal area of the hand/finger and also the time when they are able to extend the wrist.

Patients will be instructed to take their oral rescue analgesic once the pain is score >5/10.

Patients will be contacted by phone 24 hours and 48 hours after their time of arrival in PACU (time 0). They will be reminded regarding entry in the diary. They will also be asked about quality of sleep.

Patient satisfaction will be documented at 24 and 48 hours on a visual analogue scale where 0 is totally dissatisfied and 100 is totally satisfied.

The total participation time for the patients is for 2 days.

Sample size estimation The sample size is calculated for the primary outcome measure, which is the duration of the sensory block.

The duration of sensory infraclavicular block when the local anesthetic is Ropivacaine is 402 (± 183) minutes (Abdallah et al. Anesthesiology 2016; 124:683-95). With an equivalence limit (d) of 180 minutes and the calculation of the sample size with the following formula:

n = f(α, β) × 2 × σ2 / d2 (non-inferiority) and n = f(α/2, β) × 2 × σ2 / (μ1 - μ2)2 (superiority) This showed 27 patients per group (non-inferiority) and 32 patients per group (superiority), were required to ensure adequate sample size with an α of 2.5% and 95% power. We plan to have 50 patients per group, considering a high non-compliance rate.

Randomization: This will be performed using a computer generated randomization and closed envelope system. Patients will be randomized on the day of the surgical procedure. This study will be double blind because patients, anesthesiologist performing the infraclavicular block and the evaluator in the postoperative setting will not know the allocation group. The anesthesiologist providing the sedation in the Operating Room will prepare the sedative agents (Propofol and/or Dexmedetomidine) and will cover the infusions with drapes (Propofol is a white solution, the only way to hide it is to cover it with drapes). This person will not be blinded but will also not be part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male and females of 16-80 years of age, scheduled for hand, forearm and elbow ambulatory surgery with an infraclavicular block.
* American Society of Anesthesiologist (ASA) Class I, II, III
* Ability to cooperate with study related procedures

Exclusion Criteria:

* ASA IV
* Narcotic dependent (opioid intake more than 3 months) or chronic pain conditions
* Associated significant cardiac or respiratory disease, neurological deficits
* Coexisting hematological disorder or with deranged coagulation
* Pre-existing major organ dysfunction
* Psychiatric illnesses
* Emergency surgery
* Lack of informed consent
* Allergy to any of the drugs used in the study
* Surgical procedure duration greater than 3 hours

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The duration of sensory infraclavicular block in patients scheduled for upper limb surgery. | The primary outcome will be the duration of the sensory infraclavicular block in minutes, from the moment that the block is perfomed and the moment of first analgesic request.
  In the data collection form will be record the time of performance of the infraclavicular block. The patients will have a diary where they will record the time of the day when day have the first analgesic request because of pain in the surgical site.

CONTACTS AND LOCATIONS:
Overall Officials: Shalini Dhir, MD, FRCPC, Principal Investigator — Lawson Health Research Institute & Western University
Locations (1):
- Saint Joseph's Health Care London, London, Ontario, Canada